CLINICAL TRIAL: NCT05220917
Title: Comparative Effectiveness and Safety of Four Second Line Pharmacological Strategies in Type 2 Diabetes Study
Acronym: CER-4-T2D
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); VA Boston Healthcare System (U.S. Federal Agency); McGill University (Other)
Responsible Party: Principal Investigator, Elisabetta Patorno, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2021P001784
Record Dates: First submitted 2021-12-22; First posted 2022-02-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Events; Type2 Diabetes; Renal Disease
MeSH Terms: conditions — Kidney Diseases | interventions — Sodium-Glucose Transporter 2 Inhibitors; Canagliflozin; Metformin; dapagliflozin; empagliflozin; Linagliptin; Sitagliptin Phosphate; Dipeptidyl-Peptidase IV Inhibitors; Pioglitazone; Simvastatin; IDegLira; Insulin Glargine; lixisenatide; Liraglutide; dulaglutide; semaglutide; rGLP-1 protein; Exenatide; Rosiglitazone; glimepiride; Glipizide; Glyburide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (19):
- SGLT-2i (Comparison 1): For SGLT-2i vs. DPP4i SGLT-2i - exposure group DPP4i - referent group
  Interventions: Drug: SGLT2 inhibitor
- DPP-4i (Comparison 1): For SGLT-2i vs. DPP4i SGLT-2i - exposure group DPP-4i - referent group
  Interventions: Drug: DPP-4 inhibitor
- SGLT-2i (Comparison 2): For SGLT-2i vs GLP-1 RA SGLT-2i - exposure group GLP-1 RA - referent group
  Interventions: Drug: SGLT2 inhibitor
- GLP-1 RA (Comparison 2): For SGLT-2i vs GLP-1 RA SGLT-2i - exposure group GLP-1 RA - referent group
  Interventions: Drug: GLP-1RA
- GLP-1 RA (Comparison 3): For GLP-1 RA vs DPP-4i GLP-1 RA - exposure group DPP-4i - referent group
  Interventions: Drug: GLP-1RA
- DPP-4i (Comparison 3): For GLP-1 RA vs DPP-4i GLP-1 RA - exposure group DPP-4i - referent group
  Interventions: Drug: DPP-4 inhibitor
- SGLT-2i (Comparison 4): For SGLT-2i vs SU SGLT-2i - exposure group SU - referent group
  Interventions: Drug: SGLT2 inhibitor
- SU (Comparison 4): For SGLT-2i vs SU SGLT-2i - exposure group SU - referent group
  Interventions: Drug: 2nd generation SU
- GLP-1 RA (Comparison 5): For GLP-1 RA vs SU GLP-1 RA - exposure group SU - referent group
  Interventions: Drug: GLP-1RA
- SU (Comparison 5): For GLP-1 RA vs SU GLP-1 RA - exposure group SU - referent group
  Interventions: Drug: 2nd generation SU
- DPP-4i (Comparison 6): For DPP-4i vs SU DPP-4i - exposure group SU - referent group
  Interventions: Drug: DPP-4 inhibitor
- SU (Comparison 6): For DPP-4i vs SU DPP-4i - exposure group SU - referent group
  Interventions: Drug: 2nd generation SU
- SGLT2i (Comparison 7): For SGLT2i vs. GLP-1RA vs. DPP-4i vs. SU (4-way comparison) SGLT2i, GLP-1 RA, and SU - exposure groups DPP-4i - referent group
  Interventions: Drug: SGLT2 inhibitor
- GLP-1 RA (Comparison 7): For SGLT2i vs. GLP-1RA vs. DPP-4i vs. SU (4-way comparison) SGLT2i, GLP-1 RA, and SU - exposure groups DPP-4i - referent group
  Interventions: Drug: GLP-1RA
- DPP-4i (Comparison 7): For SGLT2i vs. GLP-1RA vs. DPP-4i vs. SU (4-way comparison) SGLT2i, GLP-1 RA, and SU - exposure groups DPP-4i - referent group
  Interventions: Drug: DPP-4 inhibitor
- SU (Comparison 7): For SGLT2i vs. GLP-1RA vs. DPP-4i vs. SU (4-way comparison) SGLT2i, GLP-1 RA, and SU - exposure groups DPP-4i - referent group
  Interventions: Drug: 2nd generation SU
- SGLT2i (Comparison 8): For SGLT2i vs. GLP-1RA vs. DPP-4i (3-way comparison) SGLT2i and GLP-1 RA - exposure groups DPP-4i - referent group
  Interventions: Drug: SGLT2 inhibitor
- GLP-1 RA (Comparison 8): For SGLT2i vs. GLP-1RA vs. DPP-4i (3-way comparison) SGLT2i and GLP-1 RA - exposure groups DPP-4i - referent group
  Interventions: Drug: GLP-1RA
- DPP-4i (Comparison 8): For SGLT2i vs. GLP-1RA vs. DPP-4i (3-way comparison) SGLT2i and GLP-1 RA - exposure groups DPP-4i - referent group
  Interventions: Drug: DPP-4 inhibitor

INTERVENTIONS:
Drug: SGLT2 inhibitor — Any SGLT2i dispensing claim
  Other Names: CANAGLIFLOZIN; CANAGLIFLOZIN/METFORMIN HCL; DAPAGLIFLOZIN PROPANEDIOL/METFORMIN HCL; DAPAGLIFLOZIN PROPANEDIOL; EMPAGLIFLOZIN; EMPAGLIFLOZIN/METFORMIN HCL; ERTUGLIFLOZIN PIDOLATE/METFORMIN HCL; ERTUGLIFLOZIN PIDOLATE; EMPAGLIFLOZIN/LINAGLIPTIN; EMPAGLIFLOZIN/LINAGLIPTIN/METFORMIN HCL; DAPAGLIFLOZIN PROPANEDIOL/SAXAGLIPTIN HCL; ERTUGLIFLOZIN PIDOLATE/SITAGLIPTIN PHOSPHATE
  Groups: SGLT-2i (Comparison 1); SGLT-2i (Comparison 2); SGLT-2i (Comparison 4); SGLT2i (Comparison 7); SGLT2i (Comparison 8)
Drug: DPP-4 inhibitor — Any DPP-4 inhibitor claim
  Other Names: ALOGLIPTIN BENZOATE/METFORMIN HCL; ALOGLIPTIN BENZOATE; ALOGLIPTIN BENZOATE/PIOGLITAZONE HCL; SAXAGLIPTIN HCL; SAXAGLIPTIN HCL/METFORMIN HCL; LINAGLIPTIN; LINAGLIPTIN/METFORMIN HCL; SITAGLIPTIN PHOSPHATE/METFORMIN HCL; SITAGLIPTIN PHOSPHATE; SITAGLIPTIN PHOSPHATE/SIMVASTATIN; DAPAGLIFLOZIN PROPANEDIOL/SAXAGLIPTIN HCL; EMPAGLIFLOZIN/LINAGLIPTIN; EMPAGLIFLOZIN/LINAGLIPTIN/METFORMIN HCL; ERTUGLIFLOZIN PIDOLATE/SITAGLIPTIN PHOSPHATE
  Groups: DPP-4i (Comparison 1); DPP-4i (Comparison 3); DPP-4i (Comparison 6); DPP-4i (Comparison 7); DPP-4i (Comparison 8)
Drug: GLP-1RA — Any SGLT2i dispensing claim
  Other Names: INSULIN DEGLUDEC/LIRAGLUTIDE*; INSULIN GLARGINE, HUMAN RECOMBINANT ANALOG/LIXISENATIDE*; LIXISENATIDE; LIRAGLUTIDE; DULAGLUTIDE; SEMAGLUTIDE; ALBIGLUTIDE; EXENATIDE MICROSPHERES; EXENATIDE
  Groups: GLP-1 RA (Comparison 2); GLP-1 RA (Comparison 3); GLP-1 RA (Comparison 5); GLP-1 RA (Comparison 7); GLP-1 RA (Comparison 8)
Drug: 2nd generation SU — Any 2nd generation SU claim
  Other Names: PIOGLITAZONE HCL/GLIMEPIRIDE; ROSIGLITAZONE MALEATE/GLIMEPIRIDE; GLIPIZIDE/METFORMIN HCL; GLYBURIDE,MICRONIZED; GLYBURIDE/METFORMIN HCL; GLIMEPIRIDE; GLYBURIDE; GLIPIZIDE
  Groups: SU (Comparison 4); SU (Comparison 5); SU (Comparison 6); SU (Comparison 7)

SUMMARY:
To perform an observational analysis to emulate a target trial (i.e., a hypothetical pragmatic trial that would have answered the causal question of interest) comparing the effectiveness and safety of sodium-glucose cotransporter-2 inhibitors (SGLT2i), glucagon-like peptide 1 receptor agonists (GLP-1RA), dipeptidyl peptidase-4 inhibitors (DPP-4i), and sulfonylureas (SU), at the class and individual agent level, in head-to-head comparisons in patients with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
Aim 1: (1a.) To evaluate the effectiveness of sodium-glucose cotransporter-2 inhibitors (SGLT2i), glucagon-like peptide 1 receptor agonists (GLP-1RA), dipeptidyl peptidase-4 inhibitors (DPP-4i), and sulfonylureas (SU), at the class and individual agent level, in head-to-head comparisons with respect to cardiovascular (CV) events, mortality, renal events, and other patient-centered outcomes (e.g., time spent at home), in patients with T2D and moderate baseline CV risk (event rate ≤3%/year). (1b.) To examine heterogeneity in treatment effects by age, race/ethnicity, gender, levels of CV risk, including high (≥4%/year) and low risk (<2%/year), chronic kidney disease (CKD), frailty, and multimorbidity.

Aim 2: (2a.) To monitor and quantify the association of the initiation of SGLT2i, GLP-1RA, DPP-4i, or SU, at the class and individual agent level, with previously reported drug-related harms (e.g., diabetic ketoacidosis (DKA), fractures, amputations, pancreatitis, severe hypoglycemia). (2b.) To scan study data sources for signals of potential serious unanticipated drug-related adverse events, using a data-mining approach (tree-based scan statistics). (2c.) By using data generated in Aims 2a and 2b, to build treatment-specific outcome prediction models to identify individual patients' likelihood of drug-related harms, based on specific combinations of patient features.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years for Optum Cliniformatics, IBM Marketscan, CPRD, and VHA, and ≥ 65 years for Medicare FFS at cohort entry
* At least 12 months of continuous health plan enrollment (only claims) or registration with a general practitioner (CPRD) before and including cohort entry
* Diagnosis of T2D within 12 months before (or ever before in CPRD) and including cohort entry
* Low or moderate cardiovascular (CV) risk (≤3% risk of CV events/year) at cohort entry *
* Metformin maintenance therapy, defined as 2 fills (or prescriptions in CPRD) of metformin monotherapy recorded within 6 months before and including cohort entry

Exclusion Criteria:

* Missing age or gender information
* Nursing care admission within 12 months before and including cohort entry (criteria ignored in CPRD)
* Diagnosis of type 1 diabetes within 12 months before and including cohort entry
* Diagnosis of secondary or gestational diabetes within 12 months before and including cohort entry
* Any insulin fill or prescription within 12 months before and including cohort entry
* Diagnosis of end stage renal disease (stage ≥ 5) within 12 months before and including cohort entry
* Diagnosis of acute or chronic pancreatitis within 12 months before and including cohort entry
* Diagnosis of cirrhosis or acute hepatitis within 12 months before and including cohort entry
* Diagnosis of MEN-2 within 12 months before and including cohort entry
* Recorded solid organ transplant code within 12 months before and including cohort entry
* Patients with recorded initiation of more than one agent within a comparator class at cohort entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Optum and MarketScan databases are U.S. research claims databases that include adults with employer-based health plans, with nationwide coverage for over 60 million Americans, and meaningful numbers of patients ≥65 years from Medicare Advantage plans, employer-sponsored plans covering seniors, and Medicare supplemental insurance plans. Medicare FFS is a U.S. federal health insurance program providing coverage to individuals ≥65 years and to younger individuals with disabilities. The Partners RPDR captures longitudinal EHR data for all patients that receive care at 2 large health care provider networks in the Boston metro area. The VHA is the largest integrated national health system, serving over 12 million U.S. Veterans. The VHA database includes demographic, diagnostic and procedure information from inpatient/outpatient encounters. The CPRD is comprised of two large, computerized databases of longitudinal primary care records, GOLD and Aurum, for >50 million UK patients.
Sampling Method: Non-Probability Sample
Enrollment: 781430 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
MACE | through study completion, an average of 1 year
  Myocardial Infarction, Ischemic Stroke, Cardiovascular mortality
Modified MACE | through study completion, an average of 1 year
  Myocardial Infarction, Ischemic Stroke, All-Cause mortality
Hospitalization for Heart Failure (HHF) Hospitalization for Heart Failure (HHF) | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Myocardial Infarction (MI) | through study completion, an average of 1 year
Stroke | through study completion, an average of 1 year
Cardiovascular Mortality | through study completion, an average of 1 year
All-cause mortality | through study completion, an average of 1 year
Coronary revascularization | through study completion, an average of 1 year

OTHER OUTCOMES:
CKD progression | through study completion, an average of 1 year
  Sustained decrease in eGFR, KRT (maintenance dialysis and kidney transplantation), kidney death
  * exploratory outcome, since no validated claim-based outcome definition is currently available
Sustained decrease in eGFR | through study completion, an average of 1 year
  * exploratory outcome, since no validated claim-based outcome definition is currently available
Kidney replacement therapy (KRT) | through study completion, an average of 1 year
  * exploratory outcome, since no validated claim-based outcome definition is currently available
Kidney death | through study completion, an average of 1 year
  * exploratory outcome, since no validated claim-based outcome definition is currently available
Kidney failure | through study completion, an average of 1 year
  (sustained eGFR <15 ml/min/1.73m2, maintenance dialysis and kidney transplant)
  * exploratory outcome, since no validated claim-based outcome definition is currently available
Early kidney disease | through study completion, an average of 1 year
  Defined by change in eGFR in patients with baseline eGFR > 60
  * exploratory outcome, since no validated claim-based outcome definition is currently available
Glycemic control | through study completion, an average of 1 year
  Defined by HbA1c change in patients with available baseline HbA1c
Insulin initiation | through study completion, an average of 1 year
Weight loss or gain | through study completion, an average of 1 year
  Defined by weight change in patients with available baseline weight
  * exploratory outcome, since no validated claim-based outcome definition is currently available
Diabetic ketoacidosis | through study completion, an average of 1 year
  exposure of interest - SGLT-2i
Bone fractures | through study completion, an average of 1 year
  exposure of interest - SGLT-2i
Lower-limb amputations | through study completion, an average of 1 year
  exposure of interest - SGLT-2i
Acute kidney injury | through study completion, an average of 1 year
  exposure of interest - all drug classes
Urinary infections | through study completion, an average of 1 year
  exposure of interest - SGLT-2i
Genital infections | through study completion, an average of 1 year
  exposure of interest - SGLT-2i
Acute pancreatitis | through study completion, an average of 1 year
  exposure of interest - GLP1 RA, DPP4i
Biliary events | through study completion, an average of 1 year
  exposure of interest - GLP1 RA, DPP4i
Severe hypoglycemia | through study completion, an average of 1 year
  exposure of interest - SU
Short-term retinopathy progression | through study completion, an average of 1 year
  exposure of interest - GLP1 RA
  * exploratory outcomes, since no validated outcome definition is currently available
Home time | through study completion, an average of 1 year
  Time spent out of hospital and skilled nursing facility, Time to Nursing Home Placement
Medication persistence | through study completion, an average of 1 year
  Time to discontinuation
Switching patterns | through study completion, an average of 1 year
  Treatment trajectories: patterns of use following initiation of treatment under study. To be illustrated using concentric circle diagrams or Sankey diagrams as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Patorno, MD, DrPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT05220917/Prot_SAP_001.pdf